CLINICAL TRIAL: NCT02902159
Title: Randomised Controlled Trial of an Established Direct to Public Peer Support and E-therapy Programme (Big White Wall) Versus Information to Aid Self-management of Depression and Anxiety.
Brief Title: RCT of the Effectiveness of Big White Wall Compared to Other Online Support
Acronym: REBOOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CLAHRC-EM 16053
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Depression; Anxiety
Keywords: Stress; Low Mood; Mental Health; Peer Support; Online
MeSH Terms: conditions — Depression; Anxiety Disorders; Consciousness Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BWW (Experimental): Free access to online peer support through BWW for 6 months
  Interventions: Other: BWW Online Peer Support
- MZ (Experimental): Access to NHS Moodzone Information Only
  Interventions: Other: NHS Moodzone Online Information

INTERVENTIONS:
Other: BWW Online Peer Support — Free access to BWW online peer support and other services offered by them (except live therapy), for 6 months.
  Arms: BWW
Other: NHS Moodzone Online Information — Directed to access to online information from NHS Moodzone
  Arms: MZ

SUMMARY:
A randomised controlled trial to compare the effect on wellbeing of an online peer review website (Big White Wall) compared to freely available online information (NHS Moodzone) for people with depression and anxiety.

DETAILED DESCRIPTION:
Introduction

Unipolar depression and anxiety are respectively the second and seventh leading causes of years lived with disability in the world among all health problems according to the World Health Organisation. Self-support methods of management of depression and anxiety through a population approach such as online therapy and peer support is attractive for a number of reasons including: the scale of the problem and the ability of current services to cope; providing choice about the management of their symptoms; creating personal empowerment; developing supportive social networks; recurrence prevention.

The use of public health interventions for physical conditions such as cigarette smoking, weight loss and diabetes is increasingly utilised and effective in reaching the wider public.

Big White Wall

Big White Wall (BWW) is a well-established digital service (website and apps) 3 that offers:

* Online assessment of mental health problems and physical co-morbidities
* Moderated on-line peer support
* Guided support and live therapy

It is based on public health principles, emphasises a recovery model to improve well-being and is based theoretically on a social model of depression emphasising autonomy, hopefulness and support.

There are no waiting lists, eligibility criteria and opening hours (available 24/7).

It operates a community principle that each person is supported within cultures of respect, tolerance, mutual learning and safety, and procedures such as specially trained counsellors employed by BWW as "wall guides" try to ensure that this principle is maintained.

Patterns of use are often short-term over 3 to 6 weeks but people often utilise BWW at times of further need with a substantial proportion using it for longer periods on a more regular basis. Over that time people with depression and anxiety show clinically important improvement.

The case for online peer support interventions Peer support internet interventions such as BWW take less effort for service users than internet guided cognitive behaviour therapy (CBT) as it allows the user to choose when and how to access it rather than be committed to a pre-defined course of treatment. The overall effectiveness of BWW may be in keeping with the social model of depression and anxiety from which the website was conceived; that the onset of depression or anxiety may be precipitated by insufficient social support during a time of self-perceived threat to a person's well-being from a life event. Conversely, relief from depression or anxiety may be found through increased social support and improved life events and security.

BWW can therefore guide its users towards appropriate psycho-social support as and when they require it, whilst retaining autonomy through making their own decisions about how to use that support.

An important aspect of BWW's public health approach is to reach out to isolated people with poor quality social support and a perceived threat to their wellbeing. It aims to provide a population based service that doesn't require a personal subscription so that the most disadvantaged are able to benefit. Currently BWW has been purchased by the armed forces, some universities and 25% of Clinical Commissioning groups (CCGs) throughout England which provides free access to 98% of users.

However for a wider uptake by commissioners locally and nationally the service must be tested in a randomised controlled trial (RCT) to understand who, when and how BWW is utilised and its' clinical and cost effectiveness, compared to online information alone.

Trial Objectives To use the RE-AIM framework (Reach, Effectiveness, Adoption, Implementation including economics, Maintenance) to explore the efficacy and reach of an internet intervention (online peer support) compared to online information for people with depression and anxiety.

Use qualitative analysis to determine the engagement and experiences of the participants in the BWW arm of the study to understand the motivations for use, patterns and levels of engagement (e.g. active user versus 'lurker'), negative experiences and beliefs about efficacy and role in personal empowerment.

More specifically the trial objectives are:

1. To determine the short-term clinical effectiveness of Big White Wall (BWW) versus the National Health Service (NHS) Choices Moodzone (MZ) website on well-being (primary outcome).
2. To determine the number and representativeness of participants invited and eligible to receive BWW or the NHS Choices Moodzone website.
3. To determine the number, percent and representativeness of NHS primary care practices and organisations, secondary care mental health, community and acute trust, third sector and social care organisations that referred people to either BWW or the NHS Choices Moodzone website
4. To explore the implementation of the BWW programme including barriers and drivers to reach, effectiveness and adoption and an economic evaluation of its costs and cost effectiveness from personal, social and health care perspectives.
5. To explore the maintenance of treatment effects on well-being, depressive symptoms, anxiety symptoms, quality of life and social function over 6 months in service users
6. With Academic Helth Science Network (AHSN) East Midlands to record the take up by organisations and implementation (number, percent, representativeness in East Midlands) of BWW across the East Midlands after the trial has been completed
7. Explore user engagement and experiences of BWW through qualitative interviews and text analysis

Expected duration in the trial is 6 months.

Implementation A managed network of practice will be established ideally with representation from the mental health leads from Nottingham City and Nottinghamshire CCGs and public health together with the User consultant and a GP Knowledge Broker as well as key members of National Institute of Health Research (NIHR) MindTech and the study team. This network will ensure that both the engagement strategy and the research project itself are optimised and that important learning on implementation is collected. The results of this RE-AIM study will provide a rich database of information to inform CCGs and Health and Wellbeing Boards on who BWW and other digital mental health services might reach Access to BWW across the East Midlands will depend on commissioning decisions at a public health and primary care level. At the end of the study we will work with AHSN East Midlands and Public Health England to present these findings to Directors of Public Health and mental health leads for each CCG or consortium of CCGs, Healthwatch representatives and mental health providers in the East Midlands together with a directory of alternative providers of similar services.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16+
* Live in the County of Nottinghamshire, including Nottingham City
* Scores between10-20 on the Personal Health Questionnaire (PHQ9) and/or 10+ on Genral Anxiety Disorder Scale (GAD7)
* Access to internet through a pc or smartphone (Windows, iOS, Android)
* Able and willing to give informed consent

Exclusion Criteria:

* Scores 21 or more on the PHQ-9 (severe depression)
* And /Or Scores 2 or 3 on PHQ-9 item "thoughts that you would be better off dead or of hurting yourself in some way".
* Participant does not feel that they are sufficiently proficient in the use of the English Language (BWW and Moodzone are only available in English)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Warwick-Edinburgh Mental Well-being Scale - 14 Item | 6 weeks
  Change on the 14-item Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) from baseline to week 6

SECONDARY OUTCOMES:
Warwick-Edinburgh Mental Well-being Scale - 14 Item | 12 and 26 weeks
  Maintenance of effect
Generalised Anxiety Disorder 7 Item Scale (GAD-7) | 6, 12 & 26 weeks
  Change in score on GAD7 at 6, 12 & 26 weeks
Personal Health Questionnaire 9 Item (PHQ-9) 11 | 6, 12 & 26 weeks
  Change in score at 6, 12 & 26 weeks
SF-12 v2 Health Survey 12 | 6, 12 & 26 weeks
  Change in score at 6, 12 & 26 weeks
Work and Social Adjustment Scale 8 Item - Social Function 13 | 6, 12 & 26 weeks
  Change in score at 6, 12 & 26 weeks
8-item social support measure14 | 6, 12 & 26 weeks
  Change in score at 6, 12 & 26 weeks
12-item Brugha Inventory of Life Events15 | 26 weeks
  Change in score at 26 weeks
8-item Standardised Assessment of Personality-Abbreviated Scale (SAPAS | 26 weeks
  Change in score at 6, 12 & 26 weeks

OTHER OUTCOMES:
Client Service Receipt Inventory (CSRI) | Baseline, 6, 12 & 26 weeks
  Health Economics Measure

CONTACTS AND LOCATIONS:
Overall Officials: Richard Morriss, MD, Principal Investigator — CLAHRC-EM
Locations (2):
- United Kingdom (2):
  - Nottinghamshire Healthcare NHS foundation Trust., Nottingham, Nottinghamshire
  - Nottingham University Hospitals Nhs Trust, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crisp D, Griffiths K, Mackinnon A, Bennett K, Christensen H. An online intervention for reducing depressive symptoms: secondary benefits for self-esteem, empowerment and quality of life. Psychiatry Res. 2014 Apr 30;216(1):60-6. doi: 10.1016/j.psychres.2014.01.041. Epub 2014 Feb 3. PMID 24534125
- [Background] Spiers N, Bebbington P, McManus S, Brugha TS, Jenkins R, Meltzer H. Age and birth cohort differences in the prevalence of common mental disorder in England: National Psychiatric Morbidity Surveys 1993-2007. Br J Psychiatry. 2011 Jun;198(6):479-84. doi: 10.1192/bjp.bp.110.084269. PMID 21628710
- [Background] Andrews G, Cuijpers P, Craske MG, McEvoy P, Titov N. Computer therapy for the anxiety and depressive disorders is effective, acceptable and practical health care: a meta-analysis. PLoS One. 2010 Oct 13;5(10):e13196. doi: 10.1371/journal.pone.0013196. PMID 20967242
- [Background] Gulliver A, Griffiths KM, Christensen H. Perceived barriers and facilitators to mental health help-seeking in young people: a systematic review. BMC Psychiatry. 2010 Dec 30;10:113. doi: 10.1186/1471-244X-10-113. PMID 21192795
- [Background] Mojtabai R, Olfson M, Sampson NA, Jin R, Druss B, Wang PS, Wells KB, Pincus HA, Kessler RC. Barriers to mental health treatment: results from the National Comorbidity Survey Replication. Psychol Med. 2011 Aug;41(8):1751-61. doi: 10.1017/S0033291710002291. Epub 2010 Dec 7. PMID 21134315
- [Background] Happonen AP, Kaipainen K, Vaatanen A, Kinnunen ML, Myllymaki T, Lappalainen P, Tuomela H, Rusko H, Mattila E, Lappalainen R, Korhonen I. A concept to empower self-management of psychophysiological wellbeing: preliminary user study experiences. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:312-5. doi: 10.1109/IEMBS.2009.5333549. PMID 19964215
- See also: Related Info — http://www.bigwhitewall.com